CLINICAL TRIAL: NCT01349166
Title: Effects of 3 Months of Supervised Exercise Training on Cardiometabolic and Inflammatory Biomarkers According to Glucose Tolerance (Normal, Intolerance and Type 2 Diabetes): Measures in Unstimulated and Stimulated Conditions
Brief Title: Effects of 3 Months of Supervised Exercise Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHU-0088
Record Dates: First submitted 2011-02-03; First posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Overweight/Obesity; Glucose Intolerance; Type 2 Diabetes; Sedentarity
Keywords: Obesity; Type 2 diabetes; glucose intolerance; Physical Activity; Inflammation; HPA axis; Cytokines
MeSH Terms: conditions — Overweight; Obesity; Glucose Intolerance; Diabetes Mellitus, Type 2; Motor Activity; Inflammation

INTERVENTIONS:
Behavioral: Behavior: Supervised physical training — protocol designed to evaluate effects of physical activity on cardiometabolic and inflammatory biomarkers according to glucose tolerance

SUMMARY:
The incidence of type 2 diabetes is increasing worldwide. Because of cardiovascular morbidity and mortality associated with type 2 diabetes, it is imperative to propose methods of prevention and this in early stage of abnormal glucose metabolism.

This study will assess the beneficial effects of physical activity (acute and chronic effects) (the subjects being their own controls) on cardiometabolic and inflammatory biomarkers in 3 conditions : unstimulated (fasting and resting conditions) and stimulated conditions: postprandial response to a standardized meal preceded or not by an exercise bout.

The investigators hypothesized that an acute bout of exercise will decrease the postprandial inflammatory response to a standardized meal and that this effect of exercise will be increased after 3 months of exercise training.

DETAILED DESCRIPTION:
This is a prospective study over 4 months, open, nonrandomized. 45 overweight or obese male subjects will complete 3 experimental sessions (0700-1400h) before and after 3 months of supervised physical training. During a first session, subjects will remain inactive and fasted (basal conditions). During the second session a standardized meal will be offered (postprandial response to a standardized meal). The third session will consist in the realization of an exercise bout (60min at 60%VO2 max) followed by a standardized meal (same meal that the previous day).

Several blood (catheter), salivary and urinary samples will be collected during the 3 sessions, throughout the experimental day.

ELIGIBILITY:
Inclusion Criteria:

* Male Caucasian Adults between 30 and 65 years old Sedentary criteria based on the determination of fasting glucose (WHO 1999):
* normal if fasting plasma glucose (FPG) <1.10 g / l
* diabetes if fasting glucose> 1.26 g / l (7 mmol / l) twice
* nondiabetic fasting hyperglycemia: 1.10 g / l ≤ FPG ≤ 1.26 g / l
* glucose intolerance : if plasma glucose at 120 minutes during the OGTT (75g) is between 1.40 g / l and 2 g/ l.

Body mass index 25 BMI 35kg/m2 Affiliated to National Health Insurance Subject giving his written informed consent Subject considered as normal after clinical examination and medical questionnaire

Exclusion Criteria:

* - drugs that interfere with the parameters determined
* diabetic treated with insulin, glitazones or glinides
* eating disorders like bulimia and vomiting
* special diet, vegan or vegetarian
* autoimmune disease or inflammatory progressive desease requiring prolonged treatment
* regular physical activity (> 1 hour of physical activity per week for at least 6 months)
* smoking (> 5 cigarettes / day)
* weight change greater than 5% of the total weight in the 3 months preceding the study
* contra-indication to physical activity
* chronic pathologies: cancer, inflammatory, cardiac, pulmonary, renal, gastrointestinal or liver diseases
* Being in exclusion on the National Volunteers Data file
* No one under guardianship or not subject to social security.
* Being under someone's supervision
* Subjects deprived of their liberty by judicial or administrative.
* Refusal to sign the information sheet and written consent for particip

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-08 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
supervised physical training on cardiometabolic and inflammatory biomarkers | after 3 months

SECONDARY OUTCOMES:
relationships between cortisol secretion and the postprandial inflammatory responses depending on the level of glucose tolerance | after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Principal Investigator — University Hospital, Clermont-Ferrand